CLINICAL TRIAL: NCT04354077
Title: Pilot Study to Evaluate Deep Brain Stimulation (DBS) of the Nucleus Accumbens (NAc) for Patients With Treatment-refractory Opioid Use Disorder
Brief Title: Deep Brain Stimulation Effects In Patients With Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Nestor Tomycz, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Addiction DBS
Record Dates: First submitted 2020-04-02; First posted 2020-04-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Opioid-use Disorder
Keywords: Deep Brain Stimulation; Addiction; Nucleus Accumbens
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NAc DBS (Experimental): Subjects will receive bilateral DBS of the NAc
  Interventions: Device: DBS of the NAc

INTERVENTIONS:
Device: DBS of the NAc — Deep Brain Stimulation of the Nucleus Accumbens
  Other Names: Abbott Infinity DBS lead, model 6173ANS; Abbott Infinity DBS extension, model 6371ANS; Abbott Infinity DBS implantable pulse generator, model 6660ANS; Abbott Infinity DBS guardian burr hole cap, model 6010ANS; Abbott Infinity DBS patient controller, model 6883ANS; Abbott Infinity DBS clinician programmer, model 3872ANS

SUMMARY:
This is a pilot study to evaluate the safety and efficacy of deep brain stimulation (DBS) of the nucleus accumbens (NAc) as adjunctive treatment for treatment-refractory opioid use disorder. This study will include 3 individuals with opioid use disorder and relapsing opioid use despite active participation in a drug addiction treatment program.

DETAILED DESCRIPTION:
Three (N = 3) subjects with treatment refractory opioid use disorder will receive bilateral DBS implants in the NAc using the Abbott Medical Infinity DBS system. The primary outcome of this study is to demonstrate the safety of bilateral NAc DBS in patients with treatment-refractory opioid use disorder. Secondary outcomes include time to relapse, remission of opioid use, and change in opioid craving scores. Other secondary outcomes will include the following: Hamilton Depression Scale (HDS), neurophysiological tests, body weight and biochemical markers of health and nutrition. If effective, DBS may reduce opioid use and opioid relapse in people with opioid use disorder who may continue to display relapse despite ongoing multidisciplinary standard of care. DBS brain electrode implantation and implantation of the IPGs and extension wires will be done in the operating room and will require the subject to be admitted post-operatively for an overnight stay. Two weeks after the DBS operation, subjects will undergo systematic testing each of the quadripolar contacts and formal programming. Subsequent parameter settings will be changed at routine outpatient visits based on clinical effects. Standard of care can consist of methadone or buprenorphine maintenance treatment provided by an addiction specialist.

ELIGIBILITY:
Inclusion criteria

1. Male and females age ≥ 22 years with diagnosis of opioid use disorder (OUD) based on Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) with at least a 5-year history
2. OUD must be the primary disorder
3. History of ongoing or previous opioid use, relapse, and/or cravings, despite attempts at, or attendance in, at least two different treatment modalities. These modalities may include: Comprehensive Opioid Addiction Treatment (COAT), intensive outpatient COAT, residential treatment, inpatient treatment, alternative to intensive outpatient programs, Drug Dependence Unit programs, medication-assisted treatment (MAT), medication assisted recovery (MAR), inpatient or outpatient rehabilitation, detox programs, Narcotics Anonymous, individual or group therapy, Partial Hospitalization Programs (PHP), Sober living homes, or similar interventions.
4. Self-reports ongoing opioid cravings.
5. Has completed a neuro-psychological evaluation to the satisfaction of a neuropsychologist
6. Has completed a psychiatric evaluation to the satisfaction of a psychiatrist
7. Has had a brain MRI performed and reviewed by neurosurgeon with no contraindication for DBS procedure identified
8. Platelet count > 125,000 per cubic mm and prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits
9. Negative blood cultures to rule out bacteremia

Exclusion criteria

1. Prior brain surgery
2. Baseline assessment on the Hamilton Depression Rating Scale (HAMD) of greater than 17 or moderate risk of suicide based upon a score of 3 or greater on the Columbia Suicide Severity Scale, unless clinical judgment indicates that the individual is appropriate for inclusion despite these scores.
3. History of uncontrolled or persistent seizures
4. Suspected dementia based on neuropsychological screening or Mini Mental State Exam (MMSE) Score < 25
5. Contraindications for MRI:

   1. Presence of implanted electrical stimulation device or other implanted metal devices (excluding dental braces).
   2. Claustrophobia
   3. Body weight exceeding limit of the machine (180 kg/400 lb)
6. Females who are pregnant or nursing. Female subjects of child-bearing potential must have a negative pregnancy test during the pre-op phase and must agree to utilize adequate birth control throughout the trial and for at least 30 days following trial completion.
7. Coagulopathy secondary to chronic need for anticoagulation medicine (e.g. warfarin) or anti-platelet medication (e.g. aspirin or clopidogrel)
8. Diagnosis of neurological disorders (e.g. multiple sclerosis, Parkinson's disease, and stroke)
9. Severe brain atrophy or presence of subdural hygromas or subdural hematomas on brain MRI
10. Any evidence of underlying endocarditis.
11. Primary language other than English
12. Have any other medical condition that, in the opinion of the Investigator, makes the subject unsuitable for enrollment.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Opioid use/abstinence | 6 months
  Percentage of subjects achieving opioid abstinence
Opioid use/abstinence | 1 year post-surgery
  Percentage of subjects achieving opioid abstinence

SECONDARY OUTCOMES:
Changes in biochemical markers of health | Baseline, 6, 12 and 24 months
  Biochemical battery of tests. Blood draw for plasma CBC, lytes, BUN, creatinine, Glutamate dehydrogenase (GLDH), gamma-glutamyltransferase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT), erythrocyte mean corpuscular volume (MCV), carbohydrate-deficient transferrin (CDT)
Changes in biochemical markers of nutrition | Baseline, 6, 12 and 24 months
  Biochemical battery of tests. Blood draw for plasma, pre-albumin, folate, B12, calcium, magnesium, iron
Depression score | Baseline, 3, 6, 9, 12 and 24 months post-surgery
  Hamilton Depression Scale: There are 17 items by which an assessor will select one cue which best characterizes the patient (0-4). All items are added up for a total score, where lower numbers are indicative of a normal score and higher numbers are indicative of worse depression.
Quality of life measure | Baseline, 3, 6, 9, 12 and 24 months post-surgery
  Flanagan QOL scale: Subjects will assign a rank score to 16 items. Rankings go from 7 to 1, where 7 is a better outcome and 1 is the worst outcome. The scale is as follows: 7=Delighted, 6=Pleased, 5=Mostly Satisfied, 4=Mixed, 3=Mostly Dissatisfied, 2=Unhappy, 1=Terrible. All rankings are totaled for a final score.

OTHER OUTCOMES:
Primary Safety Objective - Complication rates | 12 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Tomycz, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- AHN Allegheny General Hospital, Pittsburgh, Pennsylvania, United States